CLINICAL TRIAL: NCT06533579
Title: A Phase 1/2 Safety, Dose-finding, and Pharmacokinetics Study of VNX-101 Gene Therapy in Patients With Relapsed or Refractory CD19-Positive Hematologic Malignancies (SENTRY-CD19)
Brief Title: Gene Therapy for CD19-Positive Hematologic Malignancies (SENTRY-CD19)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vironexis Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VNX-101-01
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; Large B-cell Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Burkitt Lymphoma; Primary Mediastinal Large B-cell Lymphoma (PMBCL); Non Hodgkin Lymphoma; Mixed Phenotype Acute Leukemia
Keywords: CD19-positive; Leukemia; Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Leukemia, Biphenotypic, Acute; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1/Group 2/Group 3/Group 4 (Experimental)
  Interventions: Genetic: Dose Level 1, VNX-101; Genetic: Dose Level 2, VNX-101; Genetic: Dose Level 3, VNX-101; Genetic: Dose Level 4, VNX-101

INTERVENTIONS:
Genetic: Dose Level 1, VNX-101 — Adeno-associated viral vector encoding the CD3/CD19 Bi-Specific T-Cell Engager (AAV.CD3/CD19), Single IV infusion
Genetic: Dose Level 2, VNX-101 — Adeno-associated viral vector encoding the CD3/CD19 Bi-Specific T-Cell Engager (AAV.CD3/CD19), Single IV infusion
Genetic: Dose Level 3, VNX-101 — Adeno-associated viral vector encoding the CD3/CD19 Bi-Specific T-Cell Engager (AAV.CD3/CD19), Single IV infusion
Genetic: Dose Level 4, VNX-101 — Adeno-associated viral vector encoding the CD3/CD19 Bi-Specific T-Cell Engager (AAV.CD3/CD19), Single IV infusion

SUMMARY:
This is a Phase 1/2, first-in-human, open-label, dose-escalating trial designed to assess the safety and efficacy of VNX-101 in patients with relapsed or refractory CD19-positive hematologic malignancies.

DETAILED DESCRIPTION:
VNX-101 is an investigational adeno-associated virus (AAV) gene therapy developed to express a secreted anti-CD19/anti-CD3 scFv diabody (termed GP101). GP101 binds both cluster of differentiation (CD)19 and CD3, inducing T-cells to kill both benign and malignant B-cells. Following a single intravenous (IV) infusion, the vector induces the liver and key tissues to continuously secrete GP101 into the bloodstream, resulting in long-term, consistent serum levels of GP101. Potential advantages of VNX-101 over autologous CAR-T therapy include it is off-the-shelf, provides a gentle onset of action, does not require lymphodepletion chemotherapy, engages all T-cells continuously (including those freshly produced from the bone marrow), and utilizes highly efficient signaling through the native T-cell receptor.

In this 2-part study, dose-finding data from Part 1 of the study (n=~12 patients) will be used determine the dose for Part 2 in patients. Part 1 is a dose-finding PK study in adults ≥18 years old designed to determine the minimal dose that achieves target PK serum levels of GP101 at steady state (8-week timepoint) without dose-limited toxicities, defined as the recommended Part 2 dose (RP2D). Prior to VNX-101 dosing, subjects may undergo standard of care chemotherapy to meet dosing criteria. Part 2 (n=~20) will be opened following data safety monitoring board review of Part 1 data and is designed to determine the safety and pharmacokinetics (PK) of VNX-101 at the RP2D in a broader array of subjects. The age range for Part 2 will be expanded to include subjects ≥13 years old. Patients will be followed for safety and efficacy up to 5 years post VNX-101 dosing. Long-term follow-up assessments for safety will be conducted for 6 to 15 years post VNX-101 dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age: Part 1: 18-90 years of age, Part 2: 13-90 years of age
* Relapsed or refractory CD-19 positive leukemia or lymphoma as defined in the protocol
* CD19-positive expression
* AAV specified capsid total antibody <1:400
* Protocol-specified ranges for renal, liver, cardiac and pulmonary function
* Protocol-specified ranges for hematology parameters

Exclusion Criteria:

* Hepatoxicity (AST or ALT > 2x upper limit of normal)
* History of thrombotic microangiopathy or cardiomyopathy, or evidence of sensory neuropathy
* Pregnant or nursing (lactating) women
* Acute Graft versus Host Disease (GvHD): Grade 2-4 or chronic GvHD of any grade
* History of hypersensitivity to corticosteroids or history of corticosteroid-related toxicity
* Chemotherapy given within the protocol-specified discontinuation timelines

Other Inclusion/Exclusion criteria to be applied per protocol.

Ages: 13 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) and treatment-emergent serious events (TESAEs) | Change from Baseline to Year 5 post dosing

SECONDARY OUTCOMES:
Change from baseline in B-cell counts | Change from baseline to year 5 post dosing
Change baseline in immunoglobulin levels | Change from baseline to year 5 post dosing
Change baseline in antitumor activity | Change from baseline to year 5 post dosing
Proportion/duration of subjects achieving response, progression free survival, and disease free survival. | Change from baseline to year 5 post dosing

OTHER OUTCOMES:
Exploratory Measure: Change in VNX-101 gene product levels | Change from baseline to year 5 post dosing
Exploratory Measure: Change in VNX-101 vector shedding | Change from baseline to year 5 post dosing

CONTACTS AND LOCATIONS:
Overall Officials: Vironexis Clinical Trials, Study Director — Vironexis Biotherapeutics Inc.
Locations (8):
- United States (8):
  - City of Hope, Duarte, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - New York Medical College, Valhalla, New York
  - University of North Carolina at Chapel Hill/ University of North Carolina Medical Center, Chapel Hill, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - TriStar BMT, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://app.patientwing.com/campaign/ct.gov